CLINICAL TRIAL: NCT06930547
Title: Investigation of the Effectiveness of Smoking Cessation Education in Patients Registered at a Community Mental Health Center: A Randomized Controlled Trial
Brief Title: Effectiveness of Smoking Cessation Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 151605122024
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Tobacco Use Disorder; Mental Disorders; Smoking Cessation
Keywords: Tobacco Use Disorder; Mental Disorders; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Mental Disorders; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Experimental group Control group
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): This group will not receive the smoking cessation training.
- İntervention (Experimental): Smoking cessation training will be applied to this group
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — In this study, the experimental group will undergo a smoking cessation training program consisting of eight sessions over four weeks, conducted twice a week. Each session is planned to last approximately 40-45 minutes.
  During the program, before each session, the previous session will be reviewed to reinforce learning and establish continuity between sessions. Feedback will be collected to ensure engagement and comprehension. At the end of each session, a summary of the session's agenda will be provided.
  Before each session, both the experimental and control groups will be evaluated using a smoking cessation status form to assess their progress. Additionally, follow-up assessments will be conducted one month and three months after the program to test the retention of the training's effectiveness.
  Arms: İntervention

SUMMARY:
Smoking is an important psychosocial problem that concerns society. It is reported that 1.3 billion people use tobacco products in the world and approximately 6 million people lose their lives due to smoking every year. Despite the high mortality rate, smoking addiction is shown as one of the biggest preventable diseases and causes of death. Individuals with mental health problems have a much higher smoking rate than the general population. Studies show that people with severe mental disorders such as schizophrenia, bipolar disorder and major depression have a smoking rate three to four times higher than the general population. It has been reported that this high smoking rate is associated with more morbidity, mortality and increased healthcare costs in individuals with severe mental disorders.

It is reported that nurses, who spend the most time with patients and constitute the largest group of healthcare personnel, have an effective role in smoking cessation initiatives. The importance of nurses in tobacco control is emphasized in the publication titled "Nurses for a Tobacco-Free Life" by the International Council of Nursing (ICN). Although both national and international literature demonstrates that smoking is a serious problem in individuals with severe mental illness through descriptive research results, it is seen that smoking cessation intervention studies are quite limited. Randomized controlled intervention studies examining the effectiveness of smoking cessation interventions applied by nurses to individuals with severe mental illnesses could not be found in the literature. This study will be conducted to examine the effectiveness of smoking cessation education in patients registered in a community mental health center.

In light of this information, this study was planned as a randomized controlled study to examine the effectiveness of smoking cessation education in patients registered in a community mental health center. The data obtained from this study will reveal the effectiveness of smoking cessation education in individuals with severe mental illnesses and contribute to filling the gap in the literature in this area. In addition, a method for using smoking cessation education in individuals with severe mental illnesses will be presented with a high level of evidence study.

DETAILED DESCRIPTION:
Smoking is a significant psychosocial issue that affects society. The substance responsible for smoking addiction is nicotine, which has a stronger addictive potential than other psychoactive substances. Tobacco, in addition to its many physical health risks, is also a psychoactive substance that can lead to mental and behavioral disorders. It is estimated that 1.3 billion people worldwide use tobacco products, and approximately 8 million people die each year due to smoking. Despite the high mortality rate, smoking addiction is considered one of the leading preventable causes of disease and death.

Individuals with mental health disorders have significantly higher smoking rates compared to the general population. Studies indicate that people diagnosed with schizophrenia, bipolar disorder, and major depression smoke at a rate three to four times higher than the general public. This high smoking prevalence among individuals with severe mental illness is associated with increased morbidity, mortality, and higher healthcare costs. Reducing the burden of physical illness among people with mental disorders is recognized as a national priority, making smoking cessation among these individuals particularly important.

Nurses, who form the largest group among healthcare professionals and spend the most time with patients, play a crucial role in smoking cessation efforts. Nurses are expected to be actively involved in smoking prevention and cessation. International health authorities emphasize the need for nurses to be at the forefront of tobacco control efforts.

Global smoking cessation campaigns primarily target healthy individuals as part of preventive health strategies. However, special groups such as psychiatric patients should also be included in smoking cessation initiatives. Research indicates that a significant proportion of individuals with mental illness who smoke express a desire to quit. Furthermore, interventions that enhance smoking cessation success among the general population are also effective for individuals with mental health disorders. It is strongly recommended that evidence-based smoking cessation interventions be applied to individuals with mental disorders, just as they are to the general population.

Given the high prevalence of nicotine addiction among individuals with mental disorders and the preventable nature of smoking-related deaths, the importance of smoking cessation initiatives becomes evident. However, research has shown that mental health teams do not consistently implement evidence-based smoking cessation interventions. Although literature highlights the severity of smoking issues among individuals with severe mental illness, studies on smoking cessation interventions remain limited. Notably, randomized controlled trials examining the effectiveness of nurse-led smoking cessation interventions for this population are scarce.

This study aims to evaluate the effectiveness of smoking cessation education among patients registered at community mental health centers. It is expected to contribute to reducing smoking addiction, which is prevalent among individuals with mental disorders, while also raising awareness among mental health professionals, particularly nurses, about the importance of smoking cessation efforts.

ELIGIBILITY:
Inclusion Criteria:

* Being registered with TRSM (Community Mental Health Center)
* Being in the remission phase (the period after the patient's treatment is completed, with no observed active symptoms and improved insight)
* Smoking at least one cigarette per day regularly
* Being open to communication and collaboration
* Being over the age of 18
* Volunteering to participate in the study.

Exclusion Criteria:

* Not being registered with TRSM (Community Mental Health Center)
* Not being in the remission phase (presence of active symptoms or lack of improved insight)
* Smoking less than one cigarette per day
* Being unwilling or unable to communicate and collaborate effectively
* Being under the age of 18
* Not volunteering or unwilling to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Fagerström Test for Nicotine Dependence (FTND): | Pre-test before the training, Post-test immediately after the training, 1st follow-up 1 month after the training, 2nd follow-up 3 months after the 1st follow-up
  Developed in 1991 by Heatherton and colleagues (Heatherton et al., 1991), the FTND is a self-assessment scale used to evaluate individuals' risk of physical nicotine dependence, measure the level and intensity of addiction. It includes binary and four-point Likert-type questions, ranging between 0-1 and 0-3. The test consists of six questions, and the total score can range from 0 to 10 points. Based on the score, individuals are categorized as follows:
  0-2 points: "Very low dependence"
  3-4 points: "Low dependence"
  5 points: "Moderate dependence"
  6-7 points: "High dependence"
  8-10 points: "Very high dependence" (Uysal et al., 2004; Güneş Ersoy, 2019).
Self-Efficacy Scale | Pre-test before the training, Post-test immediately after the training, 1st follow-up 1 month after the training, 2nd follow-up 3 months after the 1st follow-up
  According to Karancı, the Self-Efficacy Scale (SES) was developed in 1984 by Nicki and colleagues. Based on social learning theories, the concept relates to an individual's belief in their ability to perform a desired behavior. Strengthening this belief is frequently used in smoking cessation efforts. The validity and reliability studies of the Self-Efficacy Scale were conducted by Karancı (1992). The scale consists of 25 items, and each item is rated on a 1-5 scale, with the options ranging from "Not sure at all: 1" to "Absolutely sure: 5". The total score ranges from 25 to 125. A higher score reflects a stronger belief in the ability to quit smoking. As the score increases, so does the belief in one's ability to quit smoking (Karancı, 1992).

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep ÖZTÜRK, PHD, Principal Investigator — Erzurum Technical University
Locations (1):
- Erzurum Community Mental Health Center, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No